CLINICAL TRIAL: NCT01927887
Title: Pre-Operative Nodal Staging of Thyroid Cancer Using Ultra-Small Superparamagnetic Iron Oxide Magnetic Resonance Imaging (USPIO MRI): Preliminary Study
Brief Title: Pre-Operative Nodal Staging of Thyroid Cancer Using USPIO MRI: Preliminary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mukesh Harisinghani, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-132
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Papillary Carcinoma of Thyroid Gland; Metastatic Medullary Thyroid Cancer; Follicular Thyroid Cancer Lymph Node Metastasis
Keywords: Papillary Carcinoma of Thyroid; Follicular thyroid cancer lymph node metastasis; Metastatic medullary thyroid cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary; Carcinoma, Medullary | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nanoparticle MRI (Experimental): Each subject will have one MRI scan. At the initial pre-scan visit, the subject will receive the ferumoxytol infusion. Within 48-72 hours after ferumoxytol infusion, a scan will be performed. Subjects will be imaged at Massachusetts General Hospital using commercial 3.0T imaging systems using dedicated neck coil and approved imaging protocols. The MR imaging will include conventional T1 and T2 weighted spin echo and 3 D gradient echo sequences.
  Interventions: Drug: Ferumoxytol; Device: Nanoparticle MRI

INTERVENTIONS:
Drug: Ferumoxytol — Ferumoxytol will be administered as an undiluted intravenous injection dose of 6 mg/kg body weight, up to a maximum dose of 510 mg, delivered at a rate of up to 1ml/sec. Each ml of the supplied agent contains 30 mg of elemental iron and the dose will be titrated based on patients body weight in kilograms; for example at a dose of 6 mg/kg, the dose for a 50 kg person will be 50 x 6 = 300 mg. As the vial contains 30 mg/ml, 10 cc of the dose will correspond to the required 300 mg dose.
  Other Names: iron oxide-ferumoxytol
Device: Nanoparticle MRI — Each subject will have one MRI scan. At the initial pre-scan visit, the subject will receive the ferumoxytol infusion. Within 48-72 hours after ferumoxytol infusion, a scan will be performed. Subjects will be imaged at Massachusetts General Hospital using commercial 3.0T imaging systems using dedicated neck coil and approved imaging protocols. The MR imaging will include conventional T1 and T2 weighted spin echo and 3 D gradient echo sequences.

SUMMARY:
The purpose of this research study is to see if a specific kind of MRI can identify small and otherwise undetected abnormal lymph nodes in patients with thyroid cancer who are undergoing surgery. The MRI is called Ultra-Small Superparamagnetic Iron Oxide Magnetic Resonance Imaging (USPIO MRI), and uses an experimental contrast agent (ferumoxytol), to try to identify these lymph nodes. The MRI uses magnetic waves to take images (pictures) of the body and is commonly used in medical testing.

Ferumoxytol is FDA approved as an iron replacement product for the treatment of iron deficiency anemia in adult patients with chronic kidney disease.

In this research study, the investigators want to see if Ferumoxytol will help to identify very small metastases that are not usually seen on standard MRI scans. If the use of USPIO MRI with the experimental agent ferumoxytol identifies very small metastases in lymph nodes, your surgeon may decide to remove them. After the surgery, the nodes will be stored and then analyzed to assess the ability of USPIO MRI and ferumoxytol to detect cancer in very small metastases in the lymph nodes.

DETAILED DESCRIPTION:
In this research study each participant will have the study MRI (USPIO MRI) before he/she undergoes surgery. Radiologists (doctors trained to read and understand this test) will review this study MRI. The imaging results will be compared with the pathology reports from the tissue removed during your surgery.

Before the research starts (screening):

After signing this consent form, the participant will be asked to undergo some screening tests or procedures to find out if the participant can be in the research study. These tests and procedures were done as part of regular care and would have been done even if it turns out that the participant does not take part in the research study.

* An tumor assessment by CT (Computerized Tomography) scan or thyroid US (ultrasonography) scans.
* If these tests show that the participant is eligible to participate in the research study, they will begin the study. If the participant does not meet the eligibility criteria, they will not be able to participate in this research study.
* Because women who are pregnant or nursing a baby cannot be in this research study, the participant will have a urine pregnancy test if they are a woman of child bearing potential. The participant cannot be in this research study if they are pregnant or breastfeeding.
* The investigator will also ask if the participant is allergic to iron. Because the study agent contains iron, the participant cannot be in this research study if they have this allergy.

After the screening procedures confirm that the Participant is eligible to participate in the research study:

The participant will have one research MRI scan:

On the first day, the participant will receive the contrast agent intravenously. This visit will take about 30 minutes.

Before injecting the contrast medium, the investigator will clean the skin on the participant's forearm with alcohol. Then the investigator will insert a small plastic tube (IV) into a vein in the participant's forearm. The investigator will give the participant the study agent, ferumoxytol, through the IV line. The dose of ferumoxytol and the rate of administration will not be more than the dose the FDA has approved when people who have anemia use this for iron replacement therapy. Before, during and until 30 minutes after the participant get the ferumoxytol, the investigator will monitor (watch) the participant closely for any reactions to the infusion. The participant will return to Massachusetts General Hospital, Boston MA 02114, 48-72 hours for the post contrast MRI. The participant will not receive Ferumoxytol before this MRI. This study visit will take about 45 minutes.

The participant will lie on a padded table. The table will move into a scanning machine. The space in the scanning machine is very narrow, just a bit wider than that participant's body. The participant will need to lie quietly for about 30 minutes while the images are being taken. If the participant has problems with claustrophobia (fear or discomfort in small or confined spaces), let the study doctor or a member of the staff know before enrolling in this study.

During the MRI procedure, the participant will hear loud "banging" noises. This is the sound the powerful magnets make during the test. The participant will be given earplugs to help reduce the noise. The participant will also be able to talk to the MRI technologist during the test and the technologist will be able to talk to the participant. If, during the test, the participant feels too uncomfortable to continue, let the technologist know, and the test will be stopped immediately.

If any of the participant's MRIs show unusual results that might be important for your health, the study doctor will contact the participant's primary surgeon. The participant's MRIs will be reviewed by a radiologist. They will be read and interpreted and the results will be communicated to the participant's surgeon before scheduled surgery. The MRI scan may show abnormal signals in lymph nodes that are outside the area that the surgeon normally removes and the surgeon may decide to extend the surgery to include this additional area. During the scheduled surgery, the participant's surgeon will remove the participant's thyroid and any lymph nodes that s/he believes are involved.

The surgery will be performed within 30 days of the MRIs. The imaging results will then be compared with the tissue that is removed during the surgery.

The thyroid and involved lymph nodes that were surgically removed will be evaluated by a pathologist and then stored for future assessment in case the thyroid cancer recurs in the body. This will allow the investigators to compare the kind of tumor removed at time of first surgery to the tumor that has recurred.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have either primary or recurrent PTC or MTC with nodal metastases detected through physical examination and/or standard imaging techniques.
* Subjects must be deemed eligible for resection by a surgeon who is listed as an Investigator in this study;
* Age > 18 years;
* Subjects must be willing and able to understand and sign Informed Consent.
* No uncontrolled serious medical or psychiatric illness.
* Women of childbearing potential must not be pregnant or lactating.
* Subjects will have had standard care CT, MRI, or ultrasound, and a fine-needle aspiration biopsy demonstrating PTC or MTC with nodal metastases or recurrent/persistent nodal disease in a patient with known PTC or MTC.

Exclusion Criteria:

* Subjects who have a known allergy to iron;
* Subjects who are pregnant or lactating;
* Subjects who are less than 18 year of age;
* Subjects with a counter-indication to MRI, such as the presence of metallic prostheses or implanted metal device (e.g., infusion pump, defibrillator)
* Subjects with sickle cell disease, hemoglobinopathy, hemochromatosis or other clinical conditions that may lead to iron overload.
* State a medical or scientific reason if women who are pregnant or nursing will be excluded from the study. Guidelines and procedures pertinent to this requirement are available at: http://ctep.cancer.gov/protocolDevelopment/templates_applications.htm. Suggested text is provided below and may be modified as necessary.

Pregnant women are excluded from this study because there are no studies of ferumoxytol in pregnant women. In animal studies, ferumoxytol caused decreased fetal weights and fetal malformations at maternally toxic doses of 13-15 times the human dose. It is unknown if ferumoxytol is present in human milk. Because of the potential for adverse events in nursing infants, a decision should be made whether to discontinue nursing or to avoid ferumoxytol.

- State a medical or scientific reason if participants who are cancer survivors or those who are HIV positive will be excluded from the study. The full text of the Policies, Guidelines, and Procedures pertinent to this requirement is available at http://ctep.cancer.gov/protocolDevelopment/templates_applications.htm.

Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy.

HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ferumoxytol and the propensity to have inflammatory adenopathy.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh G Harisinghani, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The proposed accrual goal for the study was to enroll 20 patients, who meet the inclusion criterion. 12 patients who met criteria were identified, enrolled and completed study as outlined in the protocol
Groups:
- Lymphotrophic Superparamagnetic Nanoparticles (LSN MRI): Each subject will have one MRI scan. At the initial pre-scan visit, the subject will receive the ferumoxytol infusion. Within 48-72 hours after ferumoxytol infusion, a scan will be performed. Subjects will be imaged at Massachusetts General Hospital using commercial 3.0T imaging systems using dedicated neck coil and approved imaging protocols.Ferumoxytol will be administered as an undiluted intravenous injection dose of 6 mg/kg body weight, up to a maximum dose of 510 mg, delivered at a rate of up to 1ml/sec.
Period: Overall Study
Arm/Group | Lymphotrophic Superparamagnetic Nanoparticles (LSN MRI)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Nanoparticle Enhanced MRI: Each subject will have one MRI scan at MGH. At the initial pre-scan visit, the subject will receive the ferumoxytol infusion. Within 48-72 hours after ferumoxytol infusion, a scan will be performed.The MR imaging will include conventional T1 and T2 weighted spin echo and 3 D gradient echo sequences.
  Ferumoxytol: Ferumoxytol will be administered as an undiluted intravenous injection dose of 6 mg/kg body weight, up to a maximum dose of 510 mg, delivered at a rate of up to 1ml/sec. Each ml of the supplied agent contains 30 mg of elemental iron and the dose will be titrated based on patients body weight in kilograms; for example at a dose of 6 mg/kg, the dose for a 50 kg person will be 50 x 6 = 300 mg. As the vial contains 30 mg/ml, 10 cc of the dose will correspond to the required 300 mg dose.
  lymphotrophic superparamagnetic nanoparticle
Arm/Group | Nanoparticle Enhanced MRI
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (10)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Parameters of Sensitivity of High Resolution Magnetic Resonance Imaging With Lymphotrophic Superparamagnetic Nanoparticles (LSN MRI)
Description: Using pathology as the gold standard the excised nodes will be correlated to histopathologic assessment and the primary efficacy parameters of LSN MRI will be determined for nodal staging
Time Frame: 2 Years
Measure: Number (95% Confidence Interval); unit: percentage of excised nodes
Groups:
- Lymphotrophic Superparamagnetic Nanoparticles (LSN MRI): Each subject will have one MRI scan. At the initial pre-scan visit, the subject will receive the ferumoxytol infusion. Within 48-72 hours after ferumoxytol infusion, a scan will be performed. The MR imaging will include conventional T1 and T2 weighted spin echo and 3 D gradient echo sequences.
  Ferumoxytol: Ferumoxytol will be administered as an undiluted intravenous injection dose of 6 mg/kg body weight, up to a maximum dose of 510 mg, delivered at a rate of up to 1ml/sec. Each ml of the supplied agent contains 30 mg of elemental iron and the dose will be titrated based on patients body weight in kilograms; for example at a dose of 6 mg/kg, the dose for a 50 kg person will be 50 x 6 = 300 mg. As the vial contains 30 mg/ml, 10 cc of the dose will correspond to the required 300 mg dose.
  lymphotrophic superparamagnetic nanoparticle
Arm/Group | Lymphotrophic Superparamagnetic Nanoparticles (LSN MRI)
Number analyzed (Participants) | 12
percentage of excised nodes | 85.5 [75.7 to 92]

2. Primary Outcome: Primary Efficacy Parameters of Specificity of High Resolution Magnetic Resonance Imaging With Lymphotrophic Superparamagnetic Nanoparticles (LSN MRI)
Description: Using pathology as the gold standard the excised nodes will be correlated to histopathologic assessment and the primary efficacy parameters of LSN MRI will be determined for nodal staging. Specificity was determined by assessing the percentage of true negative nodes using pathology as a gold standard.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of true negative nodes
Arm/Group | Nanoparticle MRI
Number analyzed (Participants) | 12
percentage of true negative nodes | 89.3 [85.4 to 92.4]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lymphotrophic Superparamagnetic Nanoparticles (LSN MRI)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes